CLINICAL TRIAL: NCT03002922
Title: Evaluation of Sunscreen During Exercise Under Conditions of Profuse Sweating
Brief Title: Evaluation of Sunscreen During Exercise Under Conditions of Profuse Sweating (821/2016)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18821
Record Dates: First submitted 2016-12-19; First posted 2016-12-26 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy subjects (Experimental): Subject will self-apply the test sunscreen formula to his/her face with the goal of applying 0.65 to 0.85 grams. Subject should sweat profusely.
  Interventions: Drug: BAY987517

INTERVENTIONS:
Drug: BAY987517 — Sunscreen formula Y65-158

SUMMARY:
To visually evaluate the retention of coverage of the Test Product(s) (TP) on the face after exercise compared to the full coverage observed prior to exercise

ELIGIBILITY:
Inclusion Criteria:

Subjects may be male or female, of an age of 18-55 years inclusive. Subjects must be capable of understanding and providing written informed consent.

Subjects must sign a written confidentiality agreement including a photography release form.

Subjects must be in good general health as judged by a specified licensed physician, who will indicate their suitability to participate in this study.

Exclusion Criteria:

Subjects must not have received or used an Investigational New Drug within the last 30 days.

Subjects must not have been active participants in another clinical or subjective TP performance study within the last 30 days unless authorized by this Sponsor. Subjects must not have a known physical or medical condition that would preclude vigorous exercise Subjects must not have a five-minute resting pulse rate greater than 80 bpm.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2017-01-28 (Actual); Study Completion 2017-01-28 (Actual)

PRIMARY OUTCOMES:
Change of face coverage post exercise compared to the full coverage observed prior to exercise (in percent) | At baseline, and post exercise (30 minutes)
  The expert grader will determine the percentage of coverage achieved by viewing the subject's face through the Skin Scanner

SECONDARY OUTCOMES:
Report of eye stinging assessed by questionnaire | Up to 30 minutes
  Subjective assessment of eye stinging (where 0=none to 4=severe)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hill Top Research, St. Petersburg, Florida, United States